CLINICAL TRIAL: NCT05919615
Title: Evaluation of Efficacy and Safety of Perioperative Tranexamic Acid During Primary Total Knee Arthroplasty: A Randomized, Clinical Trial
Brief Title: Use of Tranexamic Acid in the Total Knee Arthroplasty.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UDMS-Orthopedics-4-2023
Record Dates: First submitted 2023-04-24; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Knee Osteoarthritis; Blood Loss; Blood Transfusion
Keywords: tranexamic acid; total knee arthroplasty; blood loss; complication
MeSH Terms: conditions — Osteoarthritis, Knee; Hemorrhage | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: triple Blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intravenous tranexamic acid (Experimental): The intervention group comprised patients who went primary unilateral TKA and used two-dose intravenous tranexamic acid that was applied as follows: 10mg/kg of Tranexamic Acid in 100 Milliliters（ml) normal saline (0.9% sodium chloride), the first dose 15 minutes before the tourniquet deflation and the second dose at 180 minutes after the first dosage.
  Interventions: Drug: Tranexamic Acid 100 MG/ML
- placebo (Placebo Comparator): The control group comprised primary unilateral TKA patients who did not use TXA, just IV normal saline (0.9% sodium chloride).
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Tranexamic Acid 100 MG/ML — Tranexamic Acid: 100 MG/ML Solution for injection
  Other Names: TXA
  Arms: intravenous tranexamic acid
Drug: Normal saline — 0.9% sodium chloride normal saline
  Other Names: NS
  Arms: placebo

SUMMARY:
Tranexamic acid is a medication used to treat or prevent excessive blood loss during surgery. Previous studies have shown tranexamic acid (TXA) reduces blood loss and post-operative blood transfusion rate without significant complications. In addition, many meta-analyses have confirmed these results. This study also aims to determine how safe and effective tranexamic acid treatment is for different patients undergoing primary total knee arthroplasty.

DETAILED DESCRIPTION:
Tranexamic acid (TXA) is used to control both intraoperative (IO) and postoperative (PO) bleeding during various surgical procedures. Moreover, TXA was found to indirectly reduce post-surgery infection rates and decrease hemorrhage-related mortality in trauma patients. This study aims to determine how safe and effective tranexamic acid treatment is for patients undergoing primary total knee arthroplasty. The study is a prospective, randomized, triple-blinded, placebo-controlled study. Ninety participants were enrolled between July 2021 and September 2022 and followed up with every patient for six months.

The study was done in Damascus, Syria. Participants were randomly assigned following simple randomization procedures (computerized random numbers) to 1 of 2 groups. The allocation was put into concealed envelopes independent of the surgeon and the author, and the randomization was performed by a research fellow who was not involved in patient care. Participants who went unilateral primary TKA and did not use TXA, just IV normal saline (0.9% sodium chloride), formed the control group. In contrast, the intervention group comprised participants who went primary unilateral TKA and used two-dose intravenous tranexamic acid that was applied as follows: 10mg/kg of Tranexamic Acid in 100 Milliliters（ml) normal saline (0.9% sodium chloride), the first dose 15 minutes before the tourniquet deflation and the second dose at 180 minutes after the first dosage.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary knee osteoarthrosis who underwent unilateral primary TKA

Exclusion Criteria:

* Known allergic reaction to tranexamic acid
* Secondary arthritis (ex., Rheumatic arthritis, traumatic arthritis, septic arthritis)
* BMI less than 20 and more than 40.
* Patients having vascular or hematologic disease.
* Patients who were taking anti-coagulant medicine and couldn't stop it.
* Patients having acute or chronic renal failure.
* Patients classified as the AAA as grade four or five.
* Patients with intra-operative complications such as intra-operative fractures or vascular injuries.
* Post-traumatic and secondary knee arthritis patients.
* Revisions and complex primary cases.
* Patients with an active infection or a history of lower limp infection.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Total Blood Loss（TBL） | calculated by an equation at the 72h postoperative
  Total Blood Loss（TBL） in the perioperative period was calculated using the Gross formula, which is estimated by hitting the patients' blood volume by the difference between pre and post-operative hematocrit value divided by the initial hematocrit value
intra-operative blood loss | measured during surgery time (From the time of the surgical incision at the beginning of the operation until the time of wound closure at the end of the operation), Which equals about an hour
  the amount of lost blood intraoperatively and will be measured by calculating the increased weight of the utilized wet mops and the volume of the suction bottle after erasing the amount of the used lavage
post-operative blood loss | measured once 2 days after surgery
  the amount of lost blood postoperatively will be calculated as the output of the drain bottle
hidden blood loss | measured once 3 days after surgery
  the amount of lost blood in the tissues that were not measured intraoperatively or postoperatively and will be calculated using the difference between total blood loss and intra and post-operative blood loss

SECONDARY OUTCOMES:
Transfusion rates | from the day of surgery to the day of discharge,an expected average of 3 days
  Include The number of units of perioperative blood transfusions, both intraoperative and postoperative, throughout the patient's hospital stay.
perioperative complication | assesed if happened within month interval untill 6 months after surgery
  such as infection, VTE, etc

CONTACTS AND LOCATIONS:
Overall Officials: Jaber Ibrahim, M.D, Ph.D, Study Director — Damascus University
Locations (1):
- Damascus university, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alshryda S, Sarda P, Sukeik M, Nargol A, Blenkinsopp J, Mason JM. Tranexamic acid in total knee replacement: a systematic review and meta-analysis. J Bone Joint Surg Br. 2011 Dec;93(12):1577-85. doi: 10.1302/0301-620X.93B12.26989. PMID 22161917
- [Background] Wang H, Shen B, Zeng Y. Comparison of topical versus intravenous tranexamic acid in primary total knee arthroplasty: a meta-analysis of randomized controlled and prospective cohort trials. Knee. 2014 Dec;21(6):987-93. doi: 10.1016/j.knee.2014.09.010. Epub 2014 Oct 23. PMID 25450009
- [Background] Lin C, Qi Y, Jie L, Li HB, Zhao XC, Qin L, Jiang XQ, Zhang ZH, Ma L. Is combined topical with intravenous tranexamic acid superior than topical, intravenous tranexamic acid alone and control groups for blood loss controlling after total knee arthroplasty: A meta-analysis. Medicine (Baltimore). 2016 Dec;95(51):e5344. doi: 10.1097/MD.0000000000005344. PMID 28002321
- [Background] Cankaya D, Dasar U, Satilmis AB, Basaran SH, Akkaya M, Bozkurt M. The combined use of oral and topical tranexamic acid is a safe, efficient and low-cost method in reducing blood loss and transfusion rates in total knee arthroplasty. J Orthop Surg (Hong Kong). 2017 Jan;25(1):2309499016684725. doi: 10.1177/2309499016684725. PMID 28176599
- [Background] Benoni G, Lethagen S, Fredin H. The effect of tranexamic acid on local and plasma fibrinolysis during total knee arthroplasty. Thromb Res. 1997 Feb 1;85(3):195-206. doi: 10.1016/s0049-3848(97)00004-2. PMID 9058494
- [Background] Charoencholvanich K, Siriwattanasakul P. Tranexamic acid reduces blood loss and blood transfusion after TKA: a prospective randomized controlled trial. Clin Orthop Relat Res. 2011 Oct;469(10):2874-80. doi: 10.1007/s11999-011-1874-2. Epub 2011 Apr 22. PMID 21512813
- [Background] Nielsen CS, Jans O, Orsnes T, Foss NB, Troelsen A, Husted H. Combined Intra-Articular and Intravenous Tranexamic Acid Reduces Blood Loss in Total Knee Arthroplasty: A Randomized, Double-Blind, Placebo-Controlled Trial. J Bone Joint Surg Am. 2016 May 18;98(10):835-41. doi: 10.2106/JBJS.15.00810. PMID 27194493
- [Background] Berman AT, Geissele AE, Bosacco SJ. Blood loss with total knee arthroplasty. Clin Orthop Relat Res. 1988 Sep;(234):137-8. PMID 3409568
- [Background] Gross JB. Estimating allowable blood loss: corrected for dilution. Anesthesiology. 1983 Mar;58(3):277-80. doi: 10.1097/00000542-198303000-00016. No abstract available. PMID 6829965
- [Background] Marra F, Rosso F, Bruzzone M, Bonasia DE, Dettoni F, Rossi R. Use of tranexamic acid in total knee arthroplasty. Joints. 2017 Feb 7;4(4):202-213. doi: 10.11138/jts/2016.4.4.202. eCollection 2016 Oct-Dec. PMID 28217656
- [Background] Roy SP, Tanki UF, Dutta A, Jain SK, Nagi ON. Efficacy of intra-articular tranexamic acid in blood loss reduction following primary unilateral total knee arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2012 Dec;20(12):2494-501. doi: 10.1007/s00167-012-1942-5. Epub 2012 Mar 15. PMID 22419263